CLINICAL TRIAL: NCT04279717
Title: Latin-American Von Willebrand Disease Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Academia Nacional de Medicina (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol_3081
Record Dates: First submitted 2020-02-07; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Plasma, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with von Willbrand Disease Acquired
  Interventions: Other: Observation
- Subjects with von Willbrand Disease Congenital
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No interventions planned: treatment of patients at the discretion of the treating/responsible physician
  Groups: Subjects with von Willbrand Disease Congenital
Other: Observation — No interventions planned: treatment of patients at the discretion of the treating/responsible physician
  Groups: Subjects with von Willbrand Disease Acquired

SUMMARY:
Establish a Latin-American network of centers and professionals with the aim of:

* To register VWD patients in retrospective/prospective study, using a database, available online, common to all
* To register the bleeding history, the treatment and the events of VWD patients in the region
* To investigate the influence of VWD on quality of life

DETAILED DESCRIPTION:
von Willebrand disease (VWD) is the most common autosomal bleeding disorder, mostly inherited as dominant trait. VWD is due to deficiency/abnormality of von Willebrand factor (VWF). The prevalence of VWD is unknown, but estimated as 0.1% to 1% of the general population. Although the autosomal inheritance pattern would suggest an equal distribution of male and female patients, the disease is diagnosed in more females because of female-specific hemostatic challenges: menses, ovulation, pregnancy and childbirth. Diagnosis of VWD is made by assessing personal and family history of bleeding, physical examination and completed with specific laboratory tests.

There is limited information on the epidemiology of VWD in developing countries. Some countries in Latin America have registries of severe disease that, although it is the rarest form, carries the highest costs for regional health systems. So that the prevalence of clinical symptoms and laboratory features of the disease as well as the management of the disease in Latin America is unknown.

The present project aims to establish a network of centers and professionals with the objective to register and investigate all patients with VWD in Latin America, using a database available online common to all, to gain understanding about phenotype, genotype and management of VWD in the region.

ELIGIBILITY:
Inclusion Criteria:

* Historically lowest VWF:Ag and/or VWF:RCo and/or VWF:CB < 0.50 IU/ml and/or FVIII:C < 0.50 IU/ml
* All types of VWD
* All ages

Exclusion Criteria:

* Patient without consent to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with von Willebrand disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Register of VWD patients in Latin America | assessed up to 33 months
  Clinical presentation in hereditary/acquired VWD. Phenotype and genetic diagnosis.
Registration of the bleeding history | From date of selection until the date registration, assessed up to 33 months.
  Bleeding history is an essential component in the diagnosis of von Willebrand disease (VWD). ISTH Bleeding Assessment Tool (ISTH-BAT) is used to assist the diagnosis.
Response to Treatment: Follow up of FVIII, VWF:Ag and VWF:RCo | Until the end of the registry, an average of 33 months.
  The aim of therapy is to correct the dual hemostatic defect, due to defective platelet adhesion-aggregation and abnormal coagulation due to Factor VIII (FVIII) deficiency. The choice of treatment depends on a number of factors, including the severity of the bleed, the procedure planned, the subtype and severity of the disease and the age and morbidity of the patient. The evaluation of the response to the treatment is going to be through the measure of FVIII, vWF Antigen (VWF:Ag) and vWF ristocetin cofactor (vWF:RCo).
Adverse Events: Number of patients with bleeding events | until the end of the registry, an average of 33 months.
  Bleeding disorders and their treatment impact on patients, especially in women, can affect the everyday life of patients and their families. Measure of number of bleeding events, laboratory results such as Sodium.

SECONDARY OUTCOMES:
Pregnancy outcome: Follow up of FVIII, VWF:Ag and VWF:RCo | Through study completion, an average of 2 years
  For many women with VWD, pregnancy is a time of few bleeding problems. Women with Type 3 von Willebrand disease seem to have more frequent miscarriages, especially during the first trimester. The evaluation of the response to the treatment is going to be through the measure of FVIII, vWF Antigen (VWF:Ag) and vWF ristocetin cofactor (vWF:RCo).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR